CLINICAL TRIAL: NCT02177994
Title: Timing of Antibiotic Prophylaxis for Elective Cesarean Section: A Randomized Controlled Trial
Brief Title: Antibiotic Prophylaxis for Elective Cesarean Section
Acronym: TOAPFECSACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, AMR HELMY YEHIA, Lecturer in OB GYN, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TOAPFECSACT; AinShamsMH (Other: AinShamsMH)
Record Dates: First submitted 2014-06-27; First posted 2014-06-30 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Infection of Cesarian Section Wound Following Delivery
Keywords: Elective Cesarean Section; Antibiotic prophylaxis; Timing of Antibiotic prophylaxis; post cesarean section infection
MeSH Terms: interventions — Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A ceftriaxone after cord clamping (Experimental): 165 patients pregnant at 37weeks or more undergoing elective cesarean section randomly distributed to receive
  1 gm. ceftriaxone via l intravenous infusion single dose after cord clamping.
  Interventions: Drug: ceftriaxone 1gm for intravenous infusion
- Group B ceftriaxone before skin incision (Active Comparator): 165 patients pregnant at 37weeks or more undergoing elective cesarean section randomly distributed to receive
  1 gm. ceftriaxone vial intravenous infusion single dose 30-60 minutes before skin incision.
  Interventions: Drug: ceftriaxone 1gm for intravenous infusion

INTERVENTIONS:
Drug: ceftriaxone 1gm for intravenous infusion — Patients undergoing elective cesarean section with Gestational age 37 weeks or more. comparing the effect of administration of 1 gm ceftriaxone in elective cesarean section 30-60 min before skin incision versus after cord clamping.on post-cesarean section infection(wound infection as a primary outcome)
  Other Names: cefaxon

SUMMARY:
A randomized controlled study comparing the effect of administration of 1 gm ceftriaxone in elective cesarean section 30-60 min before skin incision versus after cord clamping.

DETAILED DESCRIPTION:
comparing the effect of administration of 1 gm ceftriaxone in elective cesarean section 30-60 min before skin incision versus after cord clamping.on post-cesarean section infection(wound infection as a primary outcome)

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cesarean section with Gestational age 37 weeks or more

Exclusion Criteria:

1. Fever greater than 38°C or maternal sepsis.
2. Cephalosporin allergy.
3. Exposure to any antibiotic agent within 1week before delivery.
4. Patents having premature rupture of membranes and acute chorioamnionitis.
5. Patients with chronic diseases (diabetes mellitus, renal disease and Cardiac disease).

3) Morbid obesity (BMI>30)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 328 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the rate of post cesarean section surgical site infection. | administration of 1gm ceftriaxone prophylaxis for elective cs and follow up surgical site infection till 40 days
  postoperative assessment of SSI. Patients will be followed up at 48-72 hours postoperative, at 7th days (skin suture removal) and at 6 weeks (contraception application).all patients will be contacted by telephone and interviewed. They will be rescheduled for a clinic visit if they reported signs and symptoms of wound infection (purulent discharge or erythema >1 cm in diameter, induration of the incision site and fever).

SECONDARY OUTCOMES:
other post cesarean section maternal and neonatal infection | follow up ofother post cesarean section maternal and neonatal infection till 40 days of delivery
  1. Maternal complications: other post cesarean section maternal complications, namely endometritis, pyrexia, urinary tract infection and complication of drug administration such as anaphylaxis.
  2. Neonatal complications: such as neonatal sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Amr AH Helmy, MD, Principal Investigator — Ain Shams Maternity Hospital
Locations (1):
- Antibiotic Prophylaxis for Elective Cesarean Section, Cairo, Egypt